CLINICAL TRIAL: NCT02874820
Title: I2PETPG - Quantification and Localisation of Imidazoline2 Binding Sites in a Group of Participants Diagnosed With Alzheimer's Disease Using 11C-BU99008: a Positron Emission Tomography Study
Brief Title: I2PETPG - Imidazoline2 Binding Sites in a Group of Participants Diagnosed With AD
Acronym: I2PETPG
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Patient recruitment issues.
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16HH3243; MR/L01307X/1 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
Keywords: Imidazoline Receptor 2; (4,5-dihydro-1H-imidazol-2-yl)-1-methyl-1H-indole; BU99008; [11C]-BU99008; Radionuclide Imaging; Molecular Imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — Idazoxan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient Group (Experimental): Baseline PET scan followed by a blocked PET scan
  Interventions: Radiation: [11C]BU99008; Drug: Idazoxan

INTERVENTIONS:
Radiation: [11C]BU99008 — Baseline and blocked scans
Drug: Idazoxan — Idazoxan dose up to 80mg

SUMMARY:
The imdazoline2 binding site (I2BS) is known to reside inside astrocytes. Changes in the numbers of I2BS in post mortem tissue has implicated them in a range of psychiatric conditions such as depression and addiction, along with neurodegenerative disorders such as Alzheimer's disease and Huntington's chorea. Preclinical studies have also demonstrated functional interactions with the opioid system, where I2BS ligands have been shown to affect tolerance to morphine and alleviate some of the morphine withdrawal syndrome in rats. Recently the I2BS and I2BS ligands have been shown to have some interesting analgesic effects in different models of pain.

The location of I2BS on astrocytic glial cells and the possibility that they may in some way regulate glial fibrillary acidic protein have led to increased interest into the role of I2BS and I2BS ligands in conditions characterised by marked gliosis. The number of I2BS has been shown to increase in Alzheimer's disease post mortem, and it has also been suggested that I2BS may be a marker for the severity and malignancy of human glioblastomas.

The lack of suitable imaging tools for the I2BS has meant that information regarding the number and distribution of I2BS in the brain has come from preclinical species and in vitro post-mortem studies. The recent development of [11C]BU99008 as a suitable PET ligand to quantify I2BS in vivo, enables the direct quantification of I2BS availability and regional distribution in the living human brain. In this study the investigators plan to utilise [11C]BU99008 to quantify the regional brain availability of I2BS in the human brain in vivo using PET.

DETAILED DESCRIPTION:
Participants with Alzheimer's Disease (AD) (up to 8) will receive up to two PET/CT scans with 11C-BU99008, a tracer alone and then a tracer scan following the administration of idazoxan. In addition, each participant will receive a structural MRI to enable anatomical registration of the PET data. These will enable the determination of the number and regional location of the I2BS in the brain of these conditions. These data will then be compared with that found in healthy human brains. In order to realise this, 11C-BU99008 scans alone and in conjunction with the mixed I2BS/α2-adrenoceptor drug idazoxan will be used. There is evidence that the I2BS have an age related increase in density. In order to be confident that any changes in the regional density and distribution of the I2BS that is seen is due to disease and not merely aging our AD participants will be age matched with the healthy participants.

Potential participants that pass an initial telephone screen will be invited to a screening visit where their eligibility to take part in the study will be determined and informed consent taken. This will be at the Imperial CRF and Imanova Ltd. The screening will consist of an interview where the study will be discussed and explained. The participants' understanding of the procedure, requirements and commitments confirmed and any questions answered before informed consent taken. In addition to this interview the participants personal details and demographics will be recorded and a psychiatric and medical history taken as well as the following:

* Semi-structured interviews/questionnaires will be completed: Mini International Neuropsychiatric Interview 5 (MINI 5), Cognitive diagnostic test for dementia (CAMCOG)
* A medical examination and blood taken for clinical laboratory testing.
* A structural MRI.
* Review of your medical history and current state of health, including questions about psychiatric symptoms and your use of prescription and non-prescription drugs, as well as your use of illegal drugs and alcohol.
* Physical examination such as measurements of blood pressure and heart rate, ECG.
* Collecting a urine sample to check for presence of drugs.
* Alcohol breath test.
* An "Allen's Test" will be performed to check the blood supply to your hand.
* Other questionnaires: Hospital Anxiety and Depression Scale (HADS), Eysenck personality (revised) (EPQ-R25), Spielberger Trait Anxiety Inventory (STAI), and MRI safety

Participants that are eligible will then be invited to take part in the study. The schedule detailed below is the preferred scenario, however it may be necessary to perform the MRI and PET/CT scans on separate days due to considerations of logistics or participant convenience. If for some reason it is necessary to cancel or suspend a scan due to technical reasons (e.g. radioligand production failure, scanner failure, etc.), the participant will be asked to return on another day to repeat the scan/day. This will only happen if they have not had the radioligand administered for that particular scan by the time the study is suspended. This will mean that for those participants the days on which each of these scans takes place may be different.

Each participant will receive up to two PET/CT scans and one MRI:

* Scanning Day; Morning (or Day 1) - structural MRI scan and baseline PET/CT scan with 11C-BU99008 alone to determine the total number of binding sites (total, PET signal).
* Scanning Day; Afternoon (or Day 2) - blocking PET/CT scan with 11C-BU99008 in combination with a single dose of idazoxan (I2BS block)

The combination of these two scans will allow the dissection of the regional contribution of the I2BS to the 11C-BU99008 specific signal, in order to get an accurate determination of the regional I2BS density.

Scanning day - The participants will arrive at Imanova's scanning facility in the Burlington Danes Building, Hammersmith Hospital in the early morning. The exact time will be determined by the logistical constraints of the productions of 11C-BU99008. On arrival, participants will be asked if they agree to carry on participating in the study and their general health and compliance to study specific restrictions assessed by interview, urine drugs of abuse screen and breathalyser (for alcohol). Once it is confirmed they are eligible to proceed, they will undergo the procedures.

The participants will be given a structural MRI scan and will then be cannulated in the radial artery and have a venous cannula inserted in the forearm or cubital veins. The arterial cannula is required for the collection of arterial blood sampling throughout the scan, to measure the concentration of the tracer in the arterial plasma for quantitative analysis of the PET signal. A venous cannula is required for the administration of 11C-BU99008. Baseline subjective (e.g. Spielberger State Anxiety Inventory (SSAI) and visual analogue scales (VAS)) and objective measures (e.g. heart rate (HR) and blood pressure (BP)) will be taken before they are prepared and positioned in the scanner for PET/CT scan 1. The scan will be up to 120 min in length, during which time HR and BP will be monitored. At the end of the scan, the participants will be removed and another set of subjective and objective measures taken. They will be given an acute dose of idazoxan (up to 80 mg; p.o.) about 120 min before the start of the PET/CT scan 2 and another round of subjective and objective measures and arterial blood samples taken as in PET/CT scan 1. At the end of the last PET/CT scan of the day, the participant will be removed from the scanner, any indwelling cannulae removed, a final round of subjective and objective measures recorded, and their fitness to be sent home assessed by the attending clinician. If the participants are scanned on separate days, this assessment of fitness to be sent home will occur after that days scanning. When they are fit to leave they will be sent home in a taxi.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 50 to 80 years
* Subjects who meet the NIA-AA core clinical criteria for probable Alzheimer's disease dementia
* Clinical Dementia Rating (CDR) score of 0.5 or more and MMSE ≥ 17
* Subjects on acetylcholinesterase inhibitor or memantine therapy for Alzheimer's disease must be on a stable dose prior to baseline
* Subjects must have partners/caregivers able to accompany them during the study visits, as well as monitor for, and report, any adverse events to the study team in the week after scanning
* Non-smoker
* Willing to comply with protocol and lifestyle restrictions
* Excellent understanding of English (for questionnaires)
* Participant is ambulant and capable of attending a PET scan visit as an outpatient.
* Participants with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 7.5.1. This criterion must be followed from after the first PET Scan until after the follow-up contact.
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test.
* Body weight ≥50 kg.

Exclusion Criteria:

* Current or past history of major psychiatric disorder
* Current or past history of substance use disorder
* Clinically significant brain injury or abnormality
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of or suffers from claustrophobia or subject feels unable to lie flat and still on their back for a period of up to 2 hours in the PET/CT scanner.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations or occupational exposure resulting in radiation exposure greater than 10 mSv over the past 3 years or greater than 10 mSv in a single year including the proposed study. Clinical exposure from which the subject receives a direct benefit is not included in these calculations.
* Previous inclusion in a research and/or medical protocol involving study medication within the last 3 months
* In the opinion of the study team they are unlikely to comply with the study protocol and restrictions that it imposes.
* Contraindications for subjects undergoing an MR scan (including but not limited to metal implants pacemakers, etc.)

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Density and distribution of Imidazoline 2 binding sites using either Total Volume of Distribution (VT) or Binding Potential (BP) | 1 year
  The primary outcome of this study will be the determination of the regional density and distribution of the I2BS in human brain of participants with a diagnosis of early AD. The output parameter used to determine this will be derived from the most appropriate PET pharmacokinetic model for this ligand in human. However, from our current study of this ligand in healthy volunteers this will probably be the Volume of distribution (Vt) derived from the 2 tissue compartment model (2TCM).

CONTACTS AND LOCATIONS:
Overall Officials: David J Nutt, MD, Principal Investigator — Director of Centre for Neuropsychopharmacology, Imperial College London
Locations (1):
- Centre for Neuropsychopharmacology; Division of Brain Sciences; Imperial College London; Burlington Danes Building; Hammersmith Hospital campus; 160 Du Cane Road, London, United Kingdom